CLINICAL TRIAL: NCT03878134
Title: Translational Development of Photon-Counting CT Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 190070; 19-CC-0070
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2022-01

CONDITIONS: Cancer; Inflammatory Disease; Vascular Diseases; Metabolic Bone Disease
Keywords: Photon Counting CT; Computed Tomography; Photon Counting Detectors
MeSH Terms: conditions — Neoplasms; Vascular Diseases; Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Enrolled patients may be scanned on the investigational Photon Counting CT scanner. Conventional images also obtained for comparison using the same scanner at the same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing conventional and Photon Counting CT scan on the investigational scanner (Experimental): 18 and older patients who undergo the conventional CT scan and the photon counting CT (PCCT) scan. Patient's images on the conventional scanner provide internal control to compare to the PCCT images.
  Interventions: Device: PHOTON COUNTING CT Scanner

INTERVENTIONS:
Device: PHOTON COUNTING CT Scanner — Enrolled patients will undergo the requested clinical diagnostic CT study on the investigational system using the standard detector, with or without IV and/or oral contrast as indicated and an limited scan of one body region using the PCCT detector. Both scans are able to be performed on the same scanner during the same examination.

SUMMARY:
Using an investigational CT scanner which uses a new type of detector to capture X-rays, (a photon counting CT detector), the goal of this experimental study is to compare conventional CT images to CT images using the photon counting detector in patients undergoing CT scans for clinically indicated reasons. The main question it aims to answer is whether the images produced using the new detectors are superior in quality. Participants will undergo the clinically indicated CT images and the photon counting detector CT images of a limited area during the same examination time.

DETAILED DESCRIPTION:
NIH develops new imaging techniques as one of its priorities for accelerating science, including methods for non-invasive patient assessments. Computed tomographic (CT) imaging is a mainstay of diagnostic imaging. The latest major technological advance is photon counting CT (PCCT) which uses a new x-ray detector that measures x-ray penetration of the body and the energy of each x-ray photon. NIH Clinical Center will use a prototype Siemens PCCT CounT systems built for clinical investigational use. The scanner can perform standard CT and PCCT imaging. In this protocol, NIH patients already enrolled in a clinical research protocol and who are referred to Radiology for diagnostic CT as part of that research may be enrolled in this study of PCCT. The diagnostic CT scan requested by their medical care team will be performed on the CounT scanner, providing the clinically indicated imaging, along with a single abbreviated PCCT exam of an organ or body part to support PCCT feasibility of the PCCT to provide better images in several small groups of patients with selected medical conditions. The data will be used to characterize quality of the PCCT images and to develop testable hypotheses and new diagnostic applications using PCCT capabilities.

Current CT systems, such as the Siemens SOMATOM Flash, have two x-ray tubes, each paired with an x-ray detector that measures total x-ray penetration of the patient and uses that information to create the images. The CounT scanner is a modified version of the Flash in which one of the two standard detectors has been replaced with a PCCT detector. The two imaging modes for the CounT scanner are (i) standard detector study as in a Flash scanner and (ii) PCCT scan. The patient scan will thus include clinically indicated radiation exposure with the standard detector and research radiation over a limited field with the PCCT detector. The CounT system is sited at the Clinical Center under a CRADA (Cooperative research and development agreement) with Siemens Medical Solutions.

Compared to current scanners, PCCT is expected to offer four major advantages:

* lower radiation dose
* greater spatial resolution
* reduced imaging noise
* x-ray energy discrimination

As a translational development protocol, all imaging studies are open-label and data may be analyzed as they are collected.

ELIGIBILITY:
* INCLUSION CRITERIA:
* NIH patients currently on an NIH research protocol who are referred to RAD&IS for CT examination as part of that research protocol
* 18 years old or greater
* Able to understand and sign informed consent

EXCLUSION CRITERIA:

* Studies that specifically require simultaneous dual source CT scan capability or where dual source CT scan is requested
* Studies ordered for an emergency indication
* Pregnant women. Subjects of child-bearing potential will undergo serum or urine pregnancy testing within 72 hours before examination. Post-menopausal and surgically sterilized subjects are automatically exempt from this testing
* Lactating women who are unable to stop breast feeding for 24 hours following the administration of contrast
* Body weight >500 lbs (227 kg) or a body circumference that prevents the study subject from lying flat in the scanner
* Patients who have undergone PCCT examination within the past year.
* Any contraindications that the research team identifies from the subject, RAD&IS CT questionnaires, and/or History and Assessment
* Employees or staff supervised by the Principal Investigator or an Associate will not be recruited to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Jones, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Symons R, Pourmorteza A, Sandfort V, Ahlman MA, Cropper T, Mallek M, Kappler S, Ulzheimer S, Mahesh M, Jones EC, Malayeri AA, Folio LR, Bluemke DA. Feasibility of Dose-reduced Chest CT with Photon-counting Detectors: Initial Results in Humans. Radiology. 2017 Dec;285(3):980-989. doi: 10.1148/radiol.2017162587. Epub 2017 Jul 28. PMID 28753389
- [Background] Pourmorteza A, Symons R, Henning A, Ulzheimer S, Bluemke DA. Dose Efficiency of Quarter-Millimeter Photon-Counting Computed Tomography: First-in-Human Results. Invest Radiol. 2018 Jun;53(6):365-372. doi: 10.1097/RLI.0000000000000463. PMID 29595753
- [Background] Pourmorteza A, Symons R, Reich DS, Bagheri M, Cork TE, Kappler S, Ulzheimer S, Bluemke DA. Photon-Counting CT of the Brain: In Vivo Human Results and Image-Quality Assessment. AJNR Am J Neuroradiol. 2017 Dec;38(12):2257-2263. doi: 10.3174/ajnr.A5402. Epub 2017 Oct 5. PMID 28982793
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-CC-0070.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients referred for diagnostic CT scan with clinical history or at risk status for conditions such as urologic cancers, lung cancers, as well as patients with conditions such as inflammatory lung or soft tissue diseases, arterial disorders of small vessels, or metabolic bone disease.
Groups:
- Patients Enrolled to Receive the Intervention PCCT CT Scan: 67 enrolled participants
  PHOTON COUNTING CT: Enrolled patients that could not undergo the requested clinical diagnostic CT study on the PCCT system using the standard detector, and the abbreviated PCCT scan as part of the examination. This occurred due to scheduling conflicts, and scanner down time failure to calibrate or other software Quality control failures. Patients received their CT exams on other conventional scanners and were removed from the protocol without the PCCT intervention.
  For patients who underwent the investigational scan, they completed the protocol immediately following the scan.
Period: Overall Study
Arm/Group | Patients Enrolled to Receive the Intervention PCCT CT Scan
Started | 67
Completed | 56
Not Completed | 11
Not completed — Scanner downtime or scheduling conflict | 11

BASELINE CHARACTERISTICS:
Population: 11 patients could not be scanned on the PCCT investigational scanner after being enrolled due to scanner downtime.
Groups:
- Patients Referred for Diagnostic CT Scans: up to 750 male or female, 18 and older patients
  PHOTON COUNTING CT: Enrolled patients will undergo the requested clinical diagnostic CT study on the PCCT system using the standard detector, with or without IV and/or oral contrast as indicated. They will also undergo a brief PCCT scan as part of the examination. The scan will thus include both clinically indicated radiation exposure with the standard detector and research radiation with the PCCT detector.
Arm/Group | Patients Referred for Diagnostic CT Scans
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Some patients were enrolled however were unable to receive the intervention of PCCT on the investigational CT scanner due to scanner downtime.
  years | 52 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were patients who were enrolled but were unable to undergo the intervention , PCCT CT scan due to scanner downtime.
  Participants
    Female | 39
    Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 52
  More than one race | 0
  Unknown or Not Reported | 2
Adults referred for diagnostic CT scan [Count of Participants; unit: Participants] — Patients must be adults over 18 years of age. referred for diagnostic CT based on order request in the EMR.
  Participants | 67

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Diagnostic Image Quality Grading of Photon Counting CT vs Conventional CT Images.
Description: Mean difference in relative image quality grading of CT images using Photon counting detectors vs. conventional detectors in group of patients with various clinical conditions. Scale name "Visual grading analysis (VGA)" . Expert radiologist observers compare the relative grades of the images from the PCCT to the grades of the same patient's reference images from conventional CT acquired at the same time. The visual grading scale incorporates technical factors in the acquisition and image display (such as contrast, noise and presence of artifacts and post processing). Grading is based on 5 point scale. 1- lowest image quality, 5- highest image quality. 5 is a better result. Scale as follows: 1 Images not usable- severe limitations for diagnostic use, 2 Limited -some loss of information, significant limitations for clinical use, 3 Adequate -moderate limitations for diagnostic use, 4 Good-minimal limitations for clinical use, 5 Excellent- no limitations for clinical diagnosis.
Time Frame: 2 years and 3 months, 27 months
Population: Patients with various conditions including cancer who underwent their routine conventional CT scan with additional PCCT images obtained for comparison.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Patients Enrolled in Protocol: Enrolled patients referred or invited who will undergo their clinically indicated diagnostic CT study on the PCCT system using the standard detector. They will also undergo a PCCT scan on the system restricted in extent to an organ or body part as part of the examination.
Arm/Group | Patients Enrolled in Protocol
Number analyzed (Participants) | 56
score on a scale | 0.947368421 (0.478877133)

ADVERSE EVENTS:
Time Frame: 24 hours unanticipated events related to the device are apparent at the time of scanning
Description: Events related to the diagnostic CT component are not reported. Unexpected incidental findings may be visible on the diagnostic scan read immediately or possibly only visible only on the PCCT research images which would be reviewed within 24 hours.
Groups:
- Patients Receiving the Intervention PCCT CT Scan: 57 participants, 56 individual patients. One patient was scanned twice. Each of the patient's scans was evaluated and counted as a participant.
  PHOTON COUNTING CT: Enrolled patients will undergo the requested clinical diagnostic CT study on the PCCT system using the standard detector, with or without IV and/or oral contrast as indicated. They will also undergo a brief PCCT scan as part of the examination. The scan will thus include both clinically indicated radiation exposure with the standard detector and research radiation with the PCCT detector.
Arm/Group | Patients Receiving the Intervention PCCT CT Scan
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

LIMITATIONS AND CAVEATS:
The PCCT detector and investigational CT scanner itself were in development at the time of the trial. The detector and scanner platform has been developed by industry since this time. These results are not predictive of the performance of the FDA approved PCCT scanner which was approved in October 2021.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT03878134/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT03878134/SAP_003.pdf
  • Informed Consent Form (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT03878134/ICF_004.pdf